CLINICAL TRIAL: NCT03431792
Title: The Intrauterine Fetoscopic Tracheal Occlusion (FETO) With Long Tail Balloon for a Treatment of Severe Congenital Diaphragmatic Hernia (CDH)
Brief Title: FETO With Long Tail Balloon for a Treatment of Severe CDH
Acronym: LongTailFETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Michael Tchirikov MD, PhD, Director of University Clinic of Obstetrics and Prenatal Medicine, Center of Fetal Surgery, Martin-Luther-Universität Halle-Wittenberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-104
Record Dates: First submitted 2018-01-24; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Severe Congenital Diaphragmatic Hernia
Keywords: CDH, FETO, fetal surgery, long tail FETO
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: Treatment of fetuses with severe CDH with an observed / expected total fetal lung volume ratio (o/e TFLV) ratio < 25% or with o/e TFLV ratio < 35% combined with herniation of the liver in thorax using the intrauterine fetoscopic tracheal occlusion (FETO) with the long tail latex balloon of 2.5 ml.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-Tail-FETO (Experimental): Fetus with severe CDH and o/e TFLV Ratio of < 25% or < 35% with liver herniation. The Long tail FETO will performed between 26 and 30 weeks of gestation.
  The MRI control will be perfirmed ar 32-34 weeks of gestation. Long Tail FETO: fetal i.m. application of 0.1 mg/kg Pancuronium, 1 µg/kg Fentanyl® and 0.01 mg/kg atropine. ("Long-Tail" Goldbal 5, 2,5 ml, BALT Extrusion, Montmorency, France). The fetoscope (Karl Storz, Tuttlingen, Germany) with a diameter of 1.3 mm, will be percutaneously inserted through a sheath into the uterus and then into the fetal trachea. The fetoscope will be removed and the balloon will be inserted under 4-D ultrasound guidance into the fetal trachea. The position of the balloon and suture will be visualized using the fetoscopy.
  The Long tail ballon will be removed by a second FETO after 34 weeks' gestation or bei the fetus itself with or without of the long tail balloon puncture with 22 gauge needle. The EXIT procedure is also possible.
  Interventions: Device: Long Tail Balloon

INTERVENTIONS:
Device: Long Tail Balloon — s. description of experimental Arm

SUMMARY:
Congenital diaphragmatic hernia (CDH) has an incidence of 1:2200 to 1:4000 newborns. The survival rate depends on the extent of the lung hypoplasia and pulmonary hypertension. In case of an observed / expected total fetal lung volume ratio (o/e TFLV) ratio of 25% or lower and herniation of the liver in thorax, the postnatal survival is estimated to be 10-25% or lower. The aim of fetoscopic tracheal balloon occlusion is to positively influence the lung growth in CDH fetuses avoiding the development of lung hypoplasia.

Some complications after sucsessfull FETO before delivery occur because of technical difficulties during the extraction of the balloon from the trachea, leading to asphyxia, worse outcome or neonatal demise. Jani et al. published 10 neonatal deaths from 210 FETO directly related to difficulties with the removal of the intratracheal balloon. The risk of emergent balloon removal was published to be very high (39%-56%).

Our new technique exploits the fetal ability to removal the intratracheal balloon which has been implanted for the treatment of severe CDH before the delivery, avoiding many risks associated with balloon extraction and a second fetoscopy.

The study will be performed on 20 fetuses with severe CDH. Before the FETO the total fetal lung volume ratio (o/e TFLV) will be measured by fetal MRI (magnetic . Only CDH fetuses with 24-32 weeks' gestation with o/e TFLV < 25% or the fetuses with o/e TFLV < 35% and liver herniation will be operated Second fetal MRI should be performed in one week after the FETO. The balloon will be extracted by the fetus itself before the delivery, after puncture with 22 gauge needle under ultrasound guiding, during second fetoscopy or using the EXIT (ex utero intrapartum Treatment). Neonatal follow up 12 months.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) has an incidence of 1:2200 to 1:4000 newborns, depending on whether stillbirths are included or not. 40 % of all CDH cases show associated malformations and chromosomal abnormalities and/or syndromes take place in 10-20%. The survival rate depends on the extent of the lung hypoplasia and pulmonary hypertension. Liver herniation into the thorax, is also a negative predictor of fetal survival. In case of an observed / expected total fetal lung volume ratio (o/e TFLV) ratio of 25% or lower and herniation of the liver in thorax, the postnatal survival is estimated to be 10-25% or lower. The aim of fetoscopic tracheal balloon occlusion is to positively influence the lung growth in CDH fetuses avoiding the development of lung hypoplasia.

A common complication of fetal surgery is the preterm premature rupture of membranes (PPROM) leading to preterm delivery. The next problem occurs because of technical difficulties during the extraction of the balloon from the trachea, leading to asphyxia, worse outcome or neonatal demise. Jani et al. published 10 neonatal deaths from 210 FETO directly related to difficulties with the removal of the intratracheal balloon. The risk of emergent balloon removal was published to be very high (39%-56%).

Our new long tail balloon exploits the fetal ability to removal the intratracheal balloon which has been implanted for the treatment of severe CDH before the delivery, avoiding many risks associated with balloon extraction and a second fetoscopy.

The study will be performed on 20 fetuses with severe CDH with total fetal lung volume ratio (o/e TFLV) < 25% or with o/e TFLV < 35% combined with liver herniation into the thorax. The lung volume will be estimated by fetal MRI. The selected fetuses with severe CDH at 24-32 weeks' gestation will be operated.

Before the Long tail FETO the 0.1 mg/kg Pancuronium, 1 µg/kg Fentanyl® and 0.01 mg/kg atropine will be applicated i.m. to the CDH fetus using 22 gauge needle under ultrasound control. The monofilament 5-0 polypropylene suture of 7 cm will be fixed to the balloon (Goldbal 5, 2,5 ml, BALT Extrusion, Montmorency, France) and the FETO will be performed. The fetoscope (Karl Storz, Tuttlingen, Germany) with a diameter of 1.3 mm will be percutaneously inserted through a sheath into the uterus and then into the fetal trachea. The fetoscope will be removed and the long tail balloon will be inserted under 4-D ultrasound guidance.The position of the balloon and suture will be controlled by fetoscopy and sonography.

Second fetal MRI should be performed in one week after the FETO. The balloon must be extracted before the delivery.

Possibilities of the Long tail extraction:

1. The fetus is able to extract the balloon from the trachea after FETO, by pulling the balloons' long tail, at the end of pregnancy;
2. by fetus itself after balloon puncture with 22 gauge needle under ultrasound guiding;
3. during second fetoscopy;
4. or using the EXIT procedure.

The CDH will be closed with / or without a patch. The follow up examinations will be performed at 6 and 12 months of age the baby.

ELIGIBILITY:
Inclusion Criteria:

* maternal age of 18-48 years
* severe CDH with MRI measured observed/expected total fetal lung volume (o/e TFLV) < 25% or < 35% in combination with a liver herniation into the thorax.

Exclusion Criteria:

* fetuses with other letal morphological abnormalities
* fetuses with chromosomal abnormalities
* severe maternal illneses

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
neonatal survival | 1 year
  survival rate

SECONDARY OUTCOMES:
pulmonary hypoplasia | 1 year
  clinical presence of pulmonary hypoplasia (yes - Grade /no)
Diaphragmatic Hernia operation | 1 year
  Patch (yes/no)
necrotizing enterocolitis | 1 year
  yes / no
neurodevelopmental impairment | 1 year
  (yes, - Grade /no)
APGAR | during the first 10 min after the delivery
  APGAR (1st/5th/10th min)
umbilical artery pH | during 10 min after the delivery
  pH measument in the umbilical artery
weight | 24hour
  weight in (g)
length | 24hour
  neonatal length in cm
Duration of O2-Ventilation (day) | 1 year
  Duration of O2-Ventilation (day)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tchirikov, MD, PhD, Principal Investigator — Germany, Center of Fetal Surgery, Martin-Luther University Halle-Wittenberg
Locations (1):
- Center of Fetal Surgery, Clinic of Obstetrics and Perinatal Medicine, Martin-Luther-University Halle-Wittenberg, Halle, Germany

IPD SHARING:
Plan to Share IPD: Yes
All patients:
  only the Nr. of the patient will be available, diagnosis, diaphragmatic hernia left or right, liver herniation, o/e total volume lung ration (%), gestational age at the Operation (long tail FETO), gestational age of the delivery, PPROM (yes/no), APGAR, art. pH, weight.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: when summary data are published
URL: https://web.uk-halle.de/index.php?id=7769

REFERENCES:
- [Background] Tchirikov M, Gatopoulos G, Strohner M, Puhl A, Steetskamp J. Two new approaches in intrauterine tracheal occlusion using an ultrathin fetoscope. Laryngoscope. 2010 Feb;120(2):394-8. doi: 10.1002/lary.20687. PMID 19950374
- [Background] Tchirikov M. Successful tracheal occlusion using ultrathin fetoscopic equipment combined with real-time three-dimensional ultrasound. Eur Surg Res. 2009;43(2):204-7. doi: 10.1159/000224146. Epub 2009 Jun 10. PMID 19521091
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113